CLINICAL TRIAL: NCT05341648
Title: Effects of Aerobic Exercise Program in Covid-19 Survivors With Post-Intensive Care Syndrome (Pics)
Brief Title: Aerobic Exercise and Covid-19 Survivors With Post-Intensive Care Syndrome (Pics)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01089 Saad Tariq
Record Dates: First submitted 2022-03-08; First posted 2022-04-22 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Post Intensive Care Syndrome
Keywords: Aerobic exercise; COVID-19 Survivors; Post Intensive Care Syndrome
MeSH Terms: conditions — COVID-19; postintensive care syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Aerobic Training for 3 days/week with 40-70% Intensity for 6 Weeks
  Interventions: Other: Aerobic Exercise Training
- Control group (Placebo Comparator): Home plan: Positioning, Breathing Exercises, Muscle Relaxation, and Flexibility exercises for 6 weeks
  Interventions: Other: Home Plan

INTERVENTIONS:
Other: Aerobic Exercise Training — Warm-up: 5 minutes Aerobic Training Treadmill/cycle ergometer Frequency:3 days a week Intensity:40-70% of HR max(Start from 40% than increment to as per patient tolerance) Total Duration:6 weeks. Duration of each session:15-30 mins. Cool-down: 5 minutes
  Arms: Experimental Group
Other: Home Plan — * Positions to ease breathlessness
  * Controlled breathing/Deep breathing*10 Reps* TD,s
  * Progressive Muscle Relaxation Exercises.
  * ROM & Flexibility Exercises. 3 days a week for 6 weeks.
  Arms: Control group

SUMMARY:
To investigate the effects of aerobic exercise program on physical activity, aerobic capacity, anxiety& depression in Covid-19 survivors discharged from Intensive Care Unit. There is evidence in the literature that post-intensive case survivors who have been mechanically ventilated will likely experience short- and medium-term consequences in the form of Post Intensive Care Syndrome (PICS).

DETAILED DESCRIPTION:
The notion that patients surviving intensive care and mechanical ventilation for several weeks can be discharged home without further medical attention is a dangerous illusion. Post-Intensive Care Syndrome and other severe conditions will require not only adequate screening but early rehabilitation and other interventions. So, this focused control trial will contribute particularly to determining the Effects of the Aerobic Exercise Program in Covid-19 Survivors with Post-Intensive Care Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo mechanical ventilation in the ICU.
* Recovered from Covid-19 & Discharged from ICU within the past 2 months.
* Hospital Anxiety and Depression Scale (HADS)>8.
* Scale≥ 2 on MRC Dyspnoea Scale.
* Subjects consenting to participate in the study.

Exclusion Criteria:

* Positive Covid-19 Test.
* COPD and other respiratory diseases.
* Pre-existing psychotic dementia-type illness.
* Acute neurologic diseases (meningitis, ischemic hemorrhagic stroke).
* Patients with chronic systemic disease.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression | 6 weeks
  Changes from baseline till 6 weeks, Assessed through Hospital Anxiety and Depression Scale (HADS): Questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Scoring is as followed:
  0-7 = Normal
  8-10 = Borderline abnormal (borderline case)
  11-21 = Abnormal (case)
6 min walk test: Distance (meters) | 6 weeks
  Changes from the baseline till the 6th week, 6 min walk test (6 MWT) was used to measure Functional capacity. It is a submaximal exercise test that can aid in assessing the functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters that an individual covers in 6 min without any support.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Allama Iqbal International Hospital & Mega Medical Complex., Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No